CLINICAL TRIAL: NCT06754800
Title: Pediatric Obstructive Sleep Apnea Diagnosis by Respiratory Polygraphy Including Hypopneas Associated with Autonomic Micro-arousals
Brief Title: Pediatric Obstructive Sleep Apnea Diagnosis by Respiratory Polygraphy
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2024PI033
Record Dates: First submitted 2024-03-15; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Sleep Apnea, Obstructive
Keywords: child; polysomnography; polygraphy; autonomic nervous system
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Polysomnography in routine care — Children performed a polysomnography in routine clinical care

SUMMARY:
Respiratory polygraphy (RP) can be used to detect obstructive sleep apnea syndrome in children (OSA) , but it underestimates the obstructive apnea-hypopnea index (OAHI) because hypopneas associated with cortical arousals are not evaluated. To compensate for this disadvantage, hypopneas linked with autonomic micro-arousals can be calculated from the drop in pulse wave amplitude (obtained dy oximetry), as increased respiratory efforts are related to autonomic nervous system activation, tachycardia, and elevated blood pressure.

The aim of this study is to compare OAHI obtained by RP alone or by RP considering hypopneas associated with autonomic micro-arousals with OAHI by polysomnography (PSG).

DETAILED DESCRIPTION:
The diagnosis of obstructive sleep apnea syndrome in children (OSA) requires to perform a polysomnography (PSG) in hospitalization with video surveillance and monitoring by a nurse to put the sensors back on the child if necessary. PSG gives the obstructive apnea-hypopnea index (OAHI) necessary for the diagnosis of OSA and to determine its severity. But PSG is difficult to perform in children, with several sensors and electrodes to install.

Respiratory polygraphy (RP) which uses only respiratory signals (without the neurophysiological signals ) can be used for the diagnosis of OSA but it underestimates OAHI because the hypopneas associated with cortical micro-arousals are not taken into account. An alternative to overcome this disadvantage is to determine the presence of autonomic micro-arousals because the increase in respiratory efforts during sleep is associated with activation of the autonomic nervous system and cardiovascular effects, such as tachycardia and an increase in blood pressure. Consequently, these respiratory efforts are associated either with autonomic activation or with cortical micro-arousal. One method to determine autonomic micro-arousals is photo-plethysmography which reflects sympathetic activation. Photoplethysmography is obtained by oximetry signal and is a non-invasive technique based on measuring the relative absorption by the blood of red light and infrared light through the finger. The pulsation of arterial blood flow through the finger arteries modulates light absorption and generates a pulse wave signal.

Autonomic micro-arousals will be calculated according to 3 algorithms: reduction of 1) 30%; 2) 40%; 3) 50% of the photoplethysmography signal compared to the baseline and the hypopneas associated with these decreases will be taken into account in the calculation of the OAHI. Consequently, 3 OAHI will be obtained by RP including hypopneas associated with autonomic micro-arousals.

The aim of this study is to compare OAHI obtained by RP considering hypopneas associated with autonomic micro-arousals with OAHI by PSG.

The hypothesis of this study is that RP by adding hypopneas associated with autonomic micro-arousals can identify OSA in children.

ELIGIBILITY:
Inclusion Criteria:

* Children with suspicion of OSA
* Interpretable polysomnography

Exclusion Criteria:

* Non-interpretable polysomnography

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 2 to 19 years adressed for a PSG in routine clinical care for suspicion of OSA by th ear-nose-throat physician, pediatric pulmonologist, sleep specialist, endocrtinologist, genetician
Sampling Method: Non-Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2024-12-22 (Estimated); Primary Completion 2024-12-28 (Estimated); Study Completion 2025-01-06 (Estimated)

PRIMARY OUTCOMES:
OAHI in RP including hypopneas associated with autonomic micro-arousals correlated with OAHI by PSG | A single night
  Value of OAHI in RP including hypopneas associated with autonomic micro-arousals obtained by 3 algorithms (3 values of OAHI) correlated with OAHI by PSG

SECONDARY OUTCOMES:
Diagnostic ability of RP including hypopneas associated with autonomic micro-arousals (obtained by the 3 algorithms) to diagnose OSA reported to PSG | A single night
  Sensitivity and specificity of the OAHI obtained by RP including hypopneas associated with autonomic micro-arousals to identify OSA in children
Diagnostic ability of RP including hypopneas associated with autonomic micro-arousals (obtained by the 3 algorithms) to diagnose moderate-severe OSA reported to PSG | A single night
  Sensitivity and specificity of the OAHI obtained by RP including hypopneas associated with autonomic micro-arousals to identify moderate-severe OSA in children
Determine the best of the 3 algorithms that better correlates with OAHI by PSG | A single night
  Comparison between the 3 correlation coefficients obtained from the correlation between value of OAHI in RP including hypopneas associated with autonomic micro-arousals obtained by 3 algorithms (3 values of OAHI) and OAHI by PSG

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grote L, Zou D, Kraiczi H, Hedner J. Finger plethysmography--a method for monitoring finger blood flow during sleep disordered breathing. Respir Physiol Neurobiol. 2003 Jul 16;136(2-3):141-52. doi: 10.1016/s1569-9048(03)00090-9. PMID 12853006
- [Background] Haba-Rubio J, Darbellay G, Herrmann FR, Frey JG, Fernandes A, Vesin JM, Thiran JP, Tschopp JM. Obstructive sleep apnea syndrome: effect of respiratory events and arousal on pulse wave amplitude measured by photoplethysmography in NREM sleep. Sleep Breath. 2005 Jun;9(2):73-81. doi: 10.1007/s11325-005-0017-y. PMID 15875228